



Development and Internal Validation of a Multivariable Risk Prediction Model for Severe Rebound Pain after Lower Limb Orthopedic Surgery involving Single-Shot Popliteal Sciatic Nerve Blocks: A Single Centre Retrospective Cohort Study

Protocol and Statistical Analysis Plan

Principal Investigator: Dr. Cynthia Yarnold, Clinical Assistant Professor

Department of Anesthesia, St. Paul's Hospital, Department of Anesthesiology, Pharmacology & Therapeutics, University of British Columbia

Co-Investigators: Dr. Stephan K. W. Schwarz, Professor & Dr. Jean

Templeton Hugill Chair in Anesthesia, Anesthesiology,

Pharmacology & Therapeutics, UBC

Department of Anesthesia, St. Paul's Hospital

Dr. Christopher Prabhakar, Clinical Assistant Professor

Anesthesiology, Pharmacology & Therapeutics, UBC

Department of Anesthesia, St. Paul's Hospital **Dr. Ron Ree**, Clinical Associate Professor

Anesthesiology, Pharmacology & Therapeutics, UBC

Department of Anesthesia, St. Paul's Hospital

Dr. Tim Ting Han Jen, Clinical Assistant Professor

Anesthesiology, Pharmacology & Therapeutics, UBC

Department of Anesthesia, St. Paul's Hospital **Dr. Janny Xue Chen Ke,** Anesthesiologist, Department of Anesthesia, St. Paul's Hospital

**Dr. Justine Denomme**, Clinical Fellow

Department of Anesthesia, St. Paul's Hospital

**Dr. Shih-Chieh Huang**, Medical Resident Department of Anesthesia, St. Paul's Hospital

Dr. Daniel I. McIsaac, Associate Professor of

Anesthesiology and Pain Medicine

Department of Anesthesiology and Pain Medicine,

University of Ottawa

Dr. Kevin Wing, Orthopedic Surgeon, Department of

Orthopedics, St. Paul's Hospital, UBC

**Primary Contact:** Nicola Edwards, Anesthesia Research Manager,

Department of Anesthesia, St. Paul's Hospital,





# **Study Description**

Rebound pain is a well-recognized phenomenon after the resolution of peripheral nerve blocks. (1–5) Severe rebound pain is prevalent after ambulatory surgery, with potential resultant increased health-care utilization and cost. (6) Risk factors for severe rebound pain may include younger age, female sex, high preoperative pain score, bone surgeries, and upper limb surgeries. (7–10) Use of tourniquet for lower limb procedures is also associated with worse postoperative pain compared to without. (11,12) Protective factors may include continuous perineural catheter, regional anesthesia adjuncts, and multimodal oral pain management prior to resolution of peripheral nerve blockade. (8,9,13–17) However, placement of continuous peripheral nerve block catheters utilizes additional health care resources; hence, a targeted approach where continuous perineural catheters are offered to patients at the highest risk of severe rebound pain could potentially offer the biggest benefit. The aim of the study is to derive and validate a multivariable prediction model for severe rebound pain after lower limb surgery involving popliteal blockade, to assist with risk stratification and shared decision making.

## **Primary Objectives**

The primary objective of the study is to derive and validate a multivariable clinical prediction model to predict the risk of severe pain after lower limb orthopedic surgeries after single-shot popliteal sciatic nerve blocks resolution.

## **Data Source**

The St. Paul's Hospital Peripheral Nerve Block (PNB) Database (in REDCap) will be used.

### **Study Sample**

Inclusion

Patients undergoing lower limb surgery who received single-shot popliteal sciatic nerve blocks (with or without other peripheral nerve blocks) at St. Paul's Hospital, Vancouver, from January 4, 2016 to November 1, 2019 will be included.

#### Exclusion

For patients who had multiple surgeries during the study period, only the first surgery within the study period will be selected. Patients who had uncontrolled pain (defined as NRS >3 and/or nursing note documentation of uncontrolled or severe pain and/or undocumented pain status) in the recovery room will also be excluded as this consists of a heterogenous group of patients who may have had failed block or experience pain from sites away from the blocked area, neither of which may be helped by continuous peripheral nerve block catheters. Patients receiving popliteal sciatic nerve catheters will be excluded.

### **Model Endpoints**

The primary endpoint is severe rebound pain, defined by transition from well-controlled pain (numerical rating scale [NRS] 3 or less or patient report of satisfactory pain control) in PACU while the block is working to severe pain (NRS pain score 7 or greater) within 48 h of block





performance. This definition is modified from that of Barry et al., as clinically we have noted some patients having sensory blocks lasting more than 24 hours with the use of adjuncts.

### **Lower Limb Candidate Predictors**

As there is currently no agreed method of classifying lower limb surgeries systematically as it pertains to postoperative pain, we reviewed the literature and consulted an orthopedic surgeon specializing in foot and ankle surgery (Dr. Kevin Wing) to categorize surgeries into a ranked list by anatomy, clinical similarity (e.g. fusion), and known risk factors of increased postoperative acute pain or rebound pain. If multiple surgeries are present, the surgery in the category that is deemed the most involved (i.e. higher ranking) will be selected as the primary surgery.

The following a-priori predictors were included:

- Patient will be assigned one main surgical type (i.e. surgery type is considered one class/categorical variable with Group 9 Soft tissue only as the reference):
  - o 1= Fusion/Osteotomy of Ankle/Hindfoot/Midfoot (10,18,19)
  - o 2= Total Ankle Replacement (18)
  - o 3= Acute Bony Trauma (18–22)
  - 4= Hallux Valgus Surgeries (18)
  - o 5= Hardware Removal (18)
  - o 6= Amputations
  - O 7= Other Ankle/Hindfoot/Midfoot bony procedure (19,23,24)
  - 8= Other Forefoot bony procedure (19,23,24)
  - $\circ$  9= Soft tissue only (8,18)
- Other surgical predictors
  - o Planned admission (Pre- or post-operatively) vs. ambulatory procedure
- Patient characteristics:
  - Age (continuous);
  - Sex (binary);
- Anesthesia-related:
  - Local anesthetic type (Long-acting only vs. mixed);
  - Dexamethasone use (Present or absent);
  - Intraoperative Anesthesia (General anesthesia as defined by need for advanced airway/Sedation/Spinal).

# Additional cohort characteristics to be reported:

- Pre-PNB neuropathy (Present or absent; Defined as "Yes" for either Pre-PNB neuropathy or diabetic neuropathy)
- o Tourniquet location (Leg versus thigh)
- Tourniquet duration
- Block performer (Attending/ Fellow/ Resident)
- Duration of sensory blockade (as defined by time from PNB performance to return of normal sensation) (Continuous variable);
- Duration of motor blockade (As defined by time from PNB performance to return of normal movement) (Continuous variable);



- O Time of day the nerve block wore off (Between 0000- 0700 / Between 0701-2359) (25,26)
- Health care practitioner contact, as defined by answering "yes" to the question of
  "Did you have to visit the emergency department, or call the surgeon or your family doctor for pain control after your nerve block wore off?".
- Highest pain score (HPS), as defined by the highest NRS pain score upon resolution of peripheral nerve blockade within 48 hours of block performance.

#### Methods

# **Data Preprocessing:**

# **Categorization of Lower Limb Surgeries**

In the database, the operations performed are entered as free texts, transposed from dictated operative reports. We created a standardized list of keywords and logic protocol to categorize the text variables into groups. Keywords (e.g., "total ankle replacement") will be used to electronically identify main surgical types (e.g., Group 2 = Total Ankle Replacement). Please see Supplementary Material for a full list of keywords and their corresponding surgical types. For patients who fit into multiple surgical types based on keywords, patients will be electronically assigned to the first group on the list. For example, if a patient received both bunionectomy and hardware removal, the patient will be assigned into Group 4= Hallux Valgus Surgery. All surgical assignments will subsequently be manually checked independently by two authors (T.T.H.J. and J.D.), and conflicts will be resolved with a third author (K.W.). To complement this manual check, Cohen's Kappa will be computed to identify the level of agreement of the classifications between the two authors (T.T.H.J. and J.D.), after their respective corrections to the main surgery type classifications.

# Missing values

Any variables with >10% missing data among observations will be excluded from the modelling stage. Any variables with <10% missing data among observations will have their missing values imputed using multiple imputation.

Since the primary variable of interest "Main surgery type" has numerous categorical levels, we intend to omit any observations that are missing a "Main surgery type" value, given the greater risk of non-convergence when attempting to impute this variable. Also, any observations with missing values in the primary outcome (rebound pain scores) will be excluded too. The remaining variables are assumed to be missing at random (MAR).

The planned method of multiple imputation will be by using multivariate imputation by chained equations (MICE). The following imputation techniques will be used to impute each variable with missing data:

"Predictive mean matching" will be used to impute the continuous variables



- Logistic regression will be used to impute the binary variables
- Multinomial logistic regression will be used to impute the nominal categorical variables

All variables (including the outcome) will contribute to imputation of the missing values. The plan of the imputation will be to generate 10 multiply imputed datasets (with an anticipated maximum of 20 iterations to achieve convergence), which will then be used to model and pool results.

#### **Cohort characteristics**

Summary statistics of outcomes and candidate predictors will be presented. Continuous variables will be presented as mean (SD) if normally distributed and median (IQR) if not normally distributed, and categorical variables will be presented as frequency (%).

# Model building

Correlations amongst candidate predictors will be explored to avoid risks of collinearity (for example, between dexamethasone use and type of intraoperative anesthesia). Amongst multiple highly correlated predictors, only one will be selected for the modeling based on clinical reasoning (e.g. one variable is more easily collected, less missing values, etc.). Additionally, potential multicollinearity within the final model will be diagnosed using variance inflation factors (VIF) of the predictors, with any values exceeding 4 warranting further investigation.

Multivariable logistic regression will be the statistical method used to construct a prediction model, with the above outlined imputation procedure applied to the data prior to modelling. The prediction model will contain the complete variable set as predictors (as outlined in the Candidate Predictors section). "Age", the only continuous predictor to be included in the model, will be modelled with a natural cubic spline (with 3 interior knots).

In addition, an exploratory prediction model will be created where a natural cubic spline (with 3 interior knots) will also be fitted for an additional predictor of "Tourniquet duration". This serves as an exploration of whether tourniquet duration plays a predictive role. However, this exploratory model could only be used postoperatively, when this information becomes available. Future database with information on predicted tourniquet duration would be needed for model update to minimize bias if this predictor were to be applied preoperatively. The primary and exploratory models will then be compared in terms of predictive performance and a likelihood ratio test will also be conducted to assess differences in goodness-of-fit.

To assess the performance of the predictive models, we will proceed with a bootstrap validation approach with 100 repetitions. At each repetition, the data will be sampled with replacement to form a bootstrap sample (with sample size equivalent to the original dataset). Multiple imputation will then be conducted on the bootstrap sample prior to modelling (using the same procedure outlined in the above "Missing values" section). After the pooled bootstrap model is created for the given bootstrap sample, performance measures (as discussed below) will be pooled across the 10 multiply imputed datasets of (1) the bootstrap sample and (2) the original



dataset. These will individually form estimates of the "training" and "test" performance, permitting us to compute the optimism of the pooled bootstrap model.

This process will be repeated for each of the repetitions, and optimism estimates will be averaged over the 100 repetitions. Lastly, an estimate of the original model performance will be computed by taking the apparent performance of the original model and subtracting the average optimism.

## Model performance measures

To assess model performance, we will use the area under the Receiver Operating Characteristic (ROC) curve (i.e., AUC) and calibration slope to evaluate the discrimination and calibration of the models, respectively. Other overall performance measures that will be computed include the Scaled Brier score and Nagelkerke's R<sup>2</sup>. Decile calibration plots will also be generated for the final prediction models to further assess calibration, with Loess-smoothed calibration curves created for each imputed dataset. Additionally, a decision curve analysis will be performed on the final prediction models.

Based on the final validated logistic regression models, a points system will be developed to approximate the contribution of the risk factors in the estimate of risk of having a severe rebound to increase clinical utility of the models. (27)

## Sample size

Calculations based on estimated sample size of 1270, and event rate of 50% are shown below.

# (8) [https://www.bmj.com/content/368/bmj.m441] (Excel spreadsheet of table below available)

| Binary outcomes | | |
|---|---|---|
| Figure 1 | Margin of error <=0.05 | |
| Criteria iii in pms | Outcome proportion -> | 0.5 |
| | Total n needed | 384.16 |
| Figure 2 | Mean absolute prediction error (MAPE) at 0.05 in predicted probabilities when applied to other targeted individuals | |
| | number of candidate variables -> | 18 |
| | Total n needed | 1013.2 |
| Figure 3 | Target shrinkage of <=10% (i.e. shrinkage factor = .9), Rsquared CS (proportion of variation explained) at least .1 | |
| Criteria i in pms | Total n needed | 716.234 |
| | See Fig 4 for notes: Rsq often .12 for binary for medical; use .5 for direct/explanatory | |
| Figure 5 | n participants required to ensure expected optimisim of <=0.05 in the apparent Rsq | |
| Criteria ii in pms | Anticipated Rsq | 0.2 |
| | Ln L null | -693.15 |
| | Max Rsq (depends on proportion) | 0.75 |





| n Outcome | 500 |
|-------------------------------------------------------------|---------|
| n total sample size (arbitrary) | 1000 |
| Shrinkage factor corresponding to optimism of <=0.05 in Rsq | 0.84211 |
| Total n needed | 420.427 |

| Estimate the overall outcome proportion with sufficient | |
|------------------------------------------------------------|---------|
| precision (<=0.05) | 384.16 |
| Target a small mean absolute prediction error (0.05) | 1013.2 |
| Target a shrinkage factor of 0.9 | 716.234 |
| Target small optimism of 0.05 in the apparent R2Nagelkerke | 420.427 |

Data will be analyzed using R (version 4.0.3). Any statistical tests will be two-sided, with significance levels of 0.05.



#### References

- 1. Muñoz-Leyva F, Cubillos J, Chin KJ. Managing rebound pain after regional anesthesia. Korean J Anesthesiol. 2020 Oct;73(5):372–83.
- 2. Kim J-H, Koh HJ, Kim DK, Lee H-J, Kwon K-H, Lee K-Y, et al. Interscalene brachial plexus bolus block versus patient-controlled interscalene indwelling catheter analgesia for the first 48 hours after arthroscopic rotator cuff repair. J Shoulder Elbow Surg. 2018 Jul;27(7):1243–50.
- 3. Ganta A, Ding D, Fisher N, Lavery J, Jain S, Tejwani NC. Continuous Infraclavicular Brachial Block Versus Single-Shot Nerve Block for Distal Radius Surgery: A Prospective Randomized Control Trial. J Orthop Trauma. 2018 Jan;32(1):22–6.
- 4. Ding DY, Manoli AI, Galos DK, Jain S, Tejwani NC. Continuous Popliteal Sciatic Nerve Block Versus Single Injection Nerve Block for Ankle Fracture Surgery: A Prospective Randomized Comparative Trial. J Orthop Trauma. 2015 Sep;29(9):393–8.
- 5. Abdallah FW, Halpern SH, Aoyama K, Brull R. Will the Real Benefits of Single-Shot Interscalene Block Please Stand Up? A Systematic Review and Meta-Analysis. Anesth Analg. 2015 May;120(5):1114–29.
- 6. Sunderland S, Yarnold CH, Head SJ, Osborn JA, Purssell A, Peel JK, et al. Regional Versus General Anesthesia and the Incidence of Unplanned Health Care Resource Utilization for Postoperative Pain After Wrist Fracture Surgery: Results From a Retrospective Quality Improvement Project. Reg Anesth Pain Med. 2016 Feb;41(1):22–7.
- 7. Sort R, Brorson S, Gögenur I, Nielsen JK, Møller AM. Rebound pain following peripheral nerve block anaesthesia in acute ankle fracture surgery: An exploratory pilot study. Acta Anaesthesiol Scand. 2019;63(3):396–402.
- 8. Barry GS, Bailey JG, Sardinha J, Brousseau P, Uppal V. Factors associated with rebound pain after peripheral nerve block for ambulatory surgery. Br J Anaesth [Internet]. 2020 Dec 31 [cited 2021 Feb 14];0(0). Available from: https://bjanaesthesia.org/article/S0007-0912(20)30914-4/abstract
- 9. Williams BA, Ibinson JW, Mangione MP, Modrak RT, Tonarelli EJ, Rakesh H, et al. Research priorities regarding multimodal peripheral nerve blocks for postoperative analgesia and anesthesia based on hospital quality data extracted from over 1,300 cases (2011-2014). Pain Med Malden Mass. 2015 Jan;16(1):7–12.
- 10. Gerbershagen HJ, Pogatzki-Zahn E, Aduckathil S, Peelen LM, Kappen TH, van Wijck AJM, et al. Procedure-specific risk factor analysis for the development of severe postoperative pain. Anesthesiology. 2014 May;120(5):1237–45.



- 11. Rai M, Mohapatra A, Radhesh, Bhandary B. Role of tourniquet in post-operative pain after total knee replacement surgery: a case control study. Int J Res Orthop. 2018 Oct 24;4(6):924–7.
- 12. Kumar N, Yadav C, Singh S, Kumar A, Vaithlingam A, Yadav S. Evaluation of pain in bilateral total knee replacement with and without tourniquet; a prospective randomized control trial. J Clin Orthop Trauma. 2015 Jun;6(2):85–8.
- 13. Williams BA, Bottegal MT, Kentor ML, Irrgang JJ, Williams JP. Rebound Pain Scores as a Function of Femoral Nerve Block Duration after Anterior Cruciate Ligament Reconstruction: Retrospective Analysis of a Prospective, Randomized Clinical Trial. Reg Anesth Pain Med. 2007;32(3):186–92.
- 14. Williams BA, Kentor ML, Vogt MT, Irrgang JJ, Bottegal MT, West RV, et al. Reduction of Verbal Pain Scores after Anterior Cruciate Ligament Reconstruction with 2-Day Continuous Femoral Nerve BlockA Randomized Clinical Trial. Anesthesiol J Am Soc Anesthesiol. 2006 Feb 1;104(2):315–27.
- 15. Ilfeld BM, Vandenborne K, Duncan PW, Sessler DI, Enneking FK, Shuster JJ, et al. Ambulatory continuous interscalene nerve blocks decrease the time to discharge readiness after total shoulder arthroplasty: a randomized, triple-masked, placebo-controlled study. Anesthesiology. 2006 Nov;105(5):999–1007.
- 16. Nicholson T, Maltenfort M, Getz C, Lazarus M, Williams G, Namdari S. Multimodal Pain Management Protocol Versus Patient Controlled Narcotic Analgesia for Postoperative Pain Control after Shoulder Arthroplasty. Arch Bone Jt Surg. 2018 May;6(3):196–202.
- 17. Holmberg A, Hassellund SS, Drægni T, Nordby A, Ottesen FS, Gulestøl A, et al. Analgesic effect of intravenous dexamethasone after volar plate surgery for distal radius fracture with brachial plexus block anaesthesia: a prospective, double-blind randomised clinical trial\*. Anaesthesia. 2020;75(11):1448–60.
- 18. Kvarda P, Hagemeijer NC, Waryasz G, Guss D, DiGiovanni CW, Johnson AH. Opioid Consumption Rate Following Foot and Ankle Surgery. Foot Ankle Int. 2019 Aug;40(8):905–13.
- 19. Saini S, McDonald EL, Shakked R, Nicholson K, Rogero R, Chapter M, et al. Prospective Evaluation of Utilization Patterns and Prescribing Guidelines of Opioid Consumption Following Orthopedic Foot and Ankle Surgery. Foot Ankle Int. 2018 Nov;39(11):1257–65.
- 20. Won SH, Chung CY, Park MS, Lee SY, Suh YS, Lee KM. Characteristics of and Factors Contributing to Immediate Postoperative Pain After Ankle Fracture Surgery. J Foot Ankle Surg Off Publ Am Coll Foot Ankle Surg. 2018 Oct;57(5):890–3.
- 21. Womble TN, Comadoll SM, Dugan AJ, Davenport DL, Ali SZ, Srinath A, et al. Is supplemental regional anesthesia associated with more complications and readmissions after



- ankle fracture surgery in the inpatient and outpatient setting? Foot Ankle Surg Off J Eur Soc Foot Ankle Surg. 2020 Aug 14;
- 22. Goldstein RY, Montero N, Jain SK, Egol KA, Tejwani NC. Efficacy of popliteal block in postoperative pain control after ankle fracture fixation: a prospective randomized study. J Orthop Trauma. 2012 Oct;26(10):557–61.
- 23. Merrill HM, Dean DM, Mottla JL, Neufeld SK, Cuttica DJ, Buchanan MM. Opioid Consumption Following Foot and Ankle Surgery. Foot Ankle Int. 2018 Jun;39(6):649–56.
- 24. Bhashyam AR, Keyser C, Miller CP, Jacobs J, Bluman E, Smith JT, et al. Prospective Evaluation of Opioid Use After Adoption of a Prescribing Guideline for Outpatient Foot and Ankle Surgery. Foot Ankle Int. 2019 Nov;40(11):1260–6.
- 25. Haimov I, Lavie P. Circadian Characteristics of Sleep Propensity Function in Healthy Elderly: A Comparison With Young Adults. Sleep. 1997 Apr 1;20(4):294–300.
- 26. Hirshkowitz M, Whiton K, Albert SM, Alessi C, Bruni O, DonCarlos L, et al. National Sleep Foundation's sleep time duration recommendations: methodology and results summary. Sleep Health. 2015 Mar 1;1(1):40–3.
- 27. Sullivan LM, Massaro JM, D'Agostino RB. Presentation of multivariate data for clinical use: The Framingham Study risk score functions. Stat Med. 2004 May 30;23(10):1631–60.